CLINICAL TRIAL: NCT02495909
Title: Childhood Schistosomiasis: a Novel Strategy Extending the Benefits/Reach of Antihelminthic Treatment
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: University of Zimbabwe (Other)
Responsible Party: Sponsor
Other Study IDs: MRCZ/A/1964
Record Dates: First submitted 2015-06-09; First posted 2015-07-13 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Schistosomiasis
Keywords: paediatric schistosomiasis; morbidity; immunology
MeSH Terms: conditions — Schistosomiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective and Hypotheses: This project has the overall objective of implementing and evaluating new approaches to reducing the current and future burden of urinary schistosomiasis in young children using the antihelminthic drug Praziquantel. The project aims to (1) determine the operational health benefits of treating schistosome infections early on re-infection and morbidity reduction, (2) determine if gut or urine microbiome structure (species diversity or abundance) is a risk factor for S. haematobium infection or morbidity, and (3) elucidate the factors and underlying mechanisms mediating the reduction/reversal of schistosome-related morbidity and resistance against infection/re-infection in young children.

DETAILED DESCRIPTION:
This study aims to refine current paediatric treatment of schistosomiasis using the drug Praziquantel (PZQ) to improve the current and future health of pre-school children and infants. Praziquantel is cheap, highly efficacious and safe, presenting a realistic opportunity of using a pre-existing tool in a modified way to benefit child health and development. The study will focus on children aged 3 to 5 years of age, comparing the impact of early vs. later treatment with PZQ on the current and future health status of the children. By killing worms PZQ stops the morbidity related to the presence of worms and eggs such as anaemia, abdominal pain, diarrhoea and blood in the urine as well as induced immune responses associated with reduced re-infection rates. Therefore the study will investigate the immediate health benefits of treating pre-school children and infants and the effects of treatment on re-infection rates.

ELIGIBILITY:
Inclusion Criteria:

1. lifelong residents of the area
2. have provided at least 2 urine and 2 stool for parasitological examination
3. have given a blood sample before and after each treatment episode
4. be negative for schistosomes, hookworm, Trichuris and Ascaris
5. have frequent contact with infective water

Exclusion Criteria:

1. clinical signs of tuberculosis or malaria
2. presenting with fever
3. have had a recent major operation, illness or vaccination
4. have previously received antihelminthic treatment
5. are infected with any helminths

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Zimbabwean pre-school children male and female
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-02-27 (Actual)

PRIMARY OUTCOMES:
Re-infection rates in children treated upon first infection compared to re-infection rates in children treated within 12 months of infection. | 12 months
  Compare re-infection rates in children treated upon first infection vs. those treated within 12 months of infection.

SECONDARY OUTCOMES:
Change in immune measures (cytokine and antibody levels) following curative treatment | 24 months from baseline
  Determine the change at 12 months post antihelminthic treatment from baseline of schistosome-specific (antibody levels) and systemic (cytokine levels) immune responses.
Compare the change in the gut and urine microbiome structure from baseline in children who become infected and compare to children who remain uninfected. | 12 months
  Determine the change at 12 months in the gut and urine microbiome from baseline in children who become infected and compare this to the change in the same period in age and sex matched children who remain uninfected.
Determine the treatment-related changes in systemic (cytokine levels) and schistosome- specific ( antibody levels) immune responses in children treated upon first infection vs. those treated within 12 months of infection. | 12 months
  Compare the magnitude of change from baseline in schistosome-specific (antibody levels) and systemic (cytokine levels) immune responses in children treated upon first infection to the magnitude of change from baseline in children treated within 12 months of infection at 6 weeks post-treatment
Reduction of morbidity (UACR and haematuria levels) levels in children treated upon first infection compared to morbidity reduction in children treated within 12 months of infection. | 12 Months
  Compare magnitude of the reduction of morbidity (UACR and haematuria levels)

CONTACTS AND LOCATIONS:
Overall Officials: Francisca Mutapi, PhD, Principal Investigator — University of Edinburgh
Locations (1):
- Prof Takafira Mduluza, Harare, Zimbabwe

IPD SHARING:
Plan to Share IPD: No
We do not have ethical permission to share data

REFERENCES:
- [Background] Mutapi F, Rujeni N, Bourke C, Mitchell K, Appleby L, Nausch N, Midzi N, Mduluza T. Schistosoma haematobium treatment in 1-5 year old children: safety and efficacy of the antihelminthic drug praziquantel. PLoS Negl Trop Dis. 2011 May;5(5):e1143. doi: 10.1371/journal.pntd.0001143. Epub 2011 May 17. PMID 21610855
- [Background] Mutapi F. Changing policy and practice in the control of pediatric schistosomiasis. Pediatrics. 2015 Mar;135(3):536-44. doi: 10.1542/peds.2014-3189. PMID 25687146
- [Background] Mduluza T, Mutapi F. Putting the treatment of paediatric schistosomiasis into context. Infect Dis Poverty. 2017 Apr 7;6(1):85. doi: 10.1186/s40249-017-0300-8. PMID 28388940